CLINICAL TRIAL: NCT02463032
Title: A Phase 2 Open Label, Multi-Center, Multinational, Randomized, Parallel Design Study Investigating The Efficacy and Safety Of GTx-024 On Metastatic or Locally Advanced ER+/AR+ Breast Cancer (BC) in Postmenopausal Women
Brief Title: Efficacy and Safety of GTx-024 in Patients With Estrogen Receptor (ER)+/Androgen Receptor (AR)+ Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G200802
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: ER+ and AR+ Breast Cancer
MeSH Terms: interventions — ostarine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GTx-024 9 mg (Experimental): Drug: GTx-024 GTx-024 softgel capsules will be administered once daily to a total dose of 9 mg
  Interventions: Drug: GTx-024
- GTx-024 18 mg (Experimental): Drug: GTx-024 GTx-024 softgel capsules will be administered once daily to a total dose of 18 mg
  Interventions: Drug: GTx-024

INTERVENTIONS:
Drug: GTx-024 — To determine whether either or both doses result in an acceptable clinical benefit rate.

SUMMARY:
The purpose of this study is to determine if GTx-024 at different dosages (9 mg or 18 mg) is effective and safe in the treatment of patients with metastatic or locally advanced Estrogen Receptor (ER)+ and Androgen Receptor (AR)+ breast cancer in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥ 18 years of age) with metastatic or recurrent locally advanced BC, not amenable to curative treatment by surgery or radiotherapy, with objective evidence of disease progression.

  * Women must have received ≥ 1 prior hormonal treatment(s) in the metastatic or adjuvant setting. If the most recent hormonal treatment was in the metastatic setting, duration of response (tumor regression or stabilization of disease) to this specific course of therapy must be ≥ 6 months. If the most recent hormonal treatment was in the adjuvant setting, duration of response (disease free) to this specific course of therapy must be ≥ 3 years
* Histological or cytological confirmation of ER+ BC as assessed by a local laboratory using slides, paraffin blocks, or paraffin sample or by medical history: ER+ (confirmed as ER expression more than or equal to 1% positive tumor nuclei)
* Human epidermal growth factor receptor 2 (HER2)-negative tumor by local laboratory testing (immunohistochemistry [IHC] 0, 1+ regardless of fluorescence in situ hybridization [FISH] ratio; IHC 2+ with FISH ratio lower than 2.0 or HER2 gene copy less than 6.0; FISH ratio of 0, indicating gene deletion, when positive and negative in situ hybridization [ISH] controls are present)
* Availability of paraffin embedded or formalin fixed tumor tissue; OR, a minimum of 10 and up to 20 slides of archived tumor tissue or new biopsy, if archived tissue is unavailable for central laboratory confirmation of AR status and molecular subtyping. Metastatic tumor tissue is preferred when possible.
* Postmenopausal women. Postmenopausal status is defined by the National Comprehensive Cancer Network as either:

  * Age ≥ 55 years and one year or more of amenorrhea
  * Age < 55 years and one year or more of amenorrhea, with an estradiol assay < 20 pg/mL
  * Age < 55 years and surgical menopause with bilateral oophorectomy a. Note: Ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LH-RH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression at the time of screening. Long term use (>6 months prior to screening) is permitted
* Radiological or clinical evidence (bone scan, computerized tomography [CT], and magnetic resonance Imaging [MRI]) of recurrence or progression within 30 days before randomization
* Subject must have either measurable disease or bone only non measurable disease, according to RECIST1.1
* Adequate organ function as shown by:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
  * Platelet count ≥ 100,000 cells/mm3
  * Hemoglobin (Hgb) ≥ 9.0 g/dL
  * Serum aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 2.5 upper limit of the normal range (ULN) (or ≤ 5 if hepatic metastases are present)
  * Total serum bilirubin ≤ 2.0 × ULN (unless the subject has documented Gilbert Syndrome)
  * Alkaline phosphatase levels ≤ 2.5 × ULN (≤ 5 × ULN in subjects with liver metastasis)
  * Serum creatinine ≤ 2.0 mg/dL or 177 µmol/L
  * International normalized ratio (INR), activated partial thromboplastin (aPTT), or partial thromboplastin time (PTT) < 1.5 × ULN (unless on anticoagulant treatment at screening)
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Subjects with bone metastases should be treated with intravenous bisphosphonates or subcutaneous denosumab (or investigator preferred standard of care) prior to and/or during the trial, unless there is a contraindication or subject intolerance to these therapies. For patients who are normocalcemic, therapy can be initiated at the time the patient initiates study drug
* Subject is able to swallow capsules
* Able and willing to give voluntary, written and signed informed consent before any screening procedure and according to local guidelines

Exclusion Criteria:

* Previously received > 1 course of chemotherapy (not including immunotherapies or targeted therapies) for the treatment of metastatic

  a. Note: Subjects may have received 1 course of chemotherapy prior to surgery for the treatment of locally advanced disease and 1 course of chemotherapy for the treatment of metastatic BC; however, if surgery could not be performed, this will count as the 1 chemotherapy course allowed prior to study
* Known hypersensitivity to any of the GTx-024 components or subjects previously received treatment with SARM
* Subjects with radiographic evidence of central nervous system (CNS) metastases as assessed by CT or MRI that are not well controlled (symptomatic or requiring control with continuous corticosteroid therapy [e.g., dexamethasone])

  a. Note: Subjects with CNS metastases are permitted to participate in the study if the CNS metastases are medically well-controlled and stable for at least 28 days after receiving local therapy (irradiation, surgery, etc.)
* Radiotherapy within 14 days prior to randomization except in case of localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture, which can then be completed within 7 days prior to randomization. Subjects must have recovered from radiotherapy toxicities prior to randomization
* Currently receiving hormone replacement therapy, unless discontinued prior to screening
* Subjects positive for Human Immunodeficiency Virus (HIV)
* Subject has a concomitant medical condition that precludes adequate study treatment compliance or assessment, or increases subject risk, in the opinion of the Investigator, such as but not limited to:

  * Myocardial infarction or arterial thromboembolic events within 6 months prior to Baseline or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease, or a QTcB (corrected according to Bazett's formula) interval > 470 msec
  * Serious uncontrolled cardiac arrhythmia grade II or higher according to NYHA
  * Uncontrolled hypertension (systolic > 150 and/or diastolic > 100 mm Hg)
  * Acute and chronic, active infectious disorders and non malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy
  * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
  * Another active cancer (excluding adequately treated basal cell carcinoma or cervical intraepithelial neoplasia [CIN]/cervical carcinoma in situ or melanoma in situ). Prior history of other cancer is allowed as long as there is no active disease within the prior 5 years
* Major surgery within 28 days before randomization
* Positive hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection at screening
* History of non-compliance to medical regimens
* Subjects unwilling to or unable to comply with the protocol
* Subject is currently receiving treatment with any agent listed on the prohibited medication list
* Treatment with any investigational product within < 4 half-lives for each individual investigational product OR 28 days prior to randomization
* Current treatment with intravenous bisphosphonate or denosumab with elevated serum calcium corrected for albumin or ionized calcium levels outside institutional normal limits at screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Overmoyer, MD, Principal Investigator — Susan Smith Center for Women's Cancers, Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - The West Clinic, PC, Memphis, Tennessee

REFERENCES:
- [Derived] Palmieri C, Linden H, Birrell SN, Wheelwright S, Lim E, Schwartzberg LS, Dwyer AR, Hickey TE, Rugo HS, Cobb P, O'Shaughnessy JA, Johnston S, Brufsky A, Tilley WD, Overmoyer B. Activity and safety of enobosarm, a novel, oral, selective androgen receptor modulator, in androgen receptor-positive, oestrogen receptor-positive, and HER2-negative advanced breast cancer (Study G200802): a randomised, open-label, multicentre, multinational, parallel design, phase 2 trial. Lancet Oncol. 2024 Mar;25(3):317-325. doi: 10.1016/S1470-2045(24)00004-4. Epub 2024 Feb 8. PMID 38342115

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GTx-024 9 mg | GTx-024 18 mg
Started | 72 | 64
Completed | 1 | 0
Not Completed | 71 | 64
Not completed — Lack of Efficacy | 61 | 50
Not completed — Death | 8 | 8
Not completed — Adverse Event | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GTx-024 9 mg | GTx-024 18 mg | Total
Number analyzed (Participants) | 72 | 64 | 136
Age, Continuous [Median (Full Range); unit: years] | 61 [35 to 83] | 62 [33 to 81] | 61 [33 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 64 | 136
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 70 | 59 | 129
  Unknown or Not Reported | 2 | 5 | 7
Androgen Receptor (AR) status positive [Count of Participants; unit: Participants] | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate, in Centrally Confirmed Androgen Receptor (AR)+ Subjects
Description: To estimate the clinical benefit rate (defined as complete response, partial response, or stable disease) according to RECIST 1.1, in subjects with estrogen receptor positive/androgen receptor positive (ER+/AR+) BC who have centrally confirmed AR+ status. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Clinical Benefit Rate (CBR)= CR + PR + SD.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | GTx-024 9 mg | GTx-024 18 mg
Number analyzed (Participants) | 50 | 52
participants | 16 | 15

2. Secondary Outcome: Clinical Benefit Rate, in Full Analysis Set
Description: To estimate the clinical benefit response rate in all subjects randomized who receive at least one dose of study medication (the FAS) regardless of AR status as determined by the central laboratory. o estimate the clinical benefit rate (defined as complete response, partial response, or stable disease) according to RECIST 1.1, in subjects with estrogen receptor positive/androgen receptor positive (ER+/AR+) BC who have centrally confirmed AR+ status. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Clinical Benefit Rate (CBR)= CR + PR + SD.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | GTx-024 9 mg | GTx-024 18 mg
Number analyzed (Participants) | 72 | 64
participants | 18 | 17

3. Secondary Outcome: Objective Response (CR + PR) in AR+ Patients
Description: as for outcome 1
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | GTx-024 9 mg | GTx-024 18 mg
Number analyzed (Participants) | 50 | 52
participants
  PR | 2 | 2
  CR | 2 | 0

4. Secondary Outcome: Best Overall Response in AR+ Patients
Description: To estimate the best overall response of GTx-024 9 mg and 18 mg
Time Frame: From treatment initiation to end of treatment
Measure: Number; unit: participants
Arm/Group | GTx-024 9 mg | GTx-024 18 mg
Number analyzed (Participants) | 50 | 52
participants
  PR | 2 | 2
  CR | 2 | 0

5. Secondary Outcome: Progression Free Survival in All Subjects
Description: To estimate the progression free survival of subjects receiving Gtx-024 9 mg and 18 mg. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Subjects were assessed up through 24 months.
Time Frame: From randomization to tumor progression or death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GTx-024 9 mg | GTx-024 18 mg
Number analyzed (Participants) | 72 | 64
months | 5.3 [NA to NA] — Due to the study ending prematurely and the limited data available, the confidence interval was not reported. This data is NOT available as it was never provided to GTx- the median was the only reported value. All good cause efforts to locate the data have been exhausted, data are missing and hence not available to be reported. | 2.9 [NA to NA] — Due to the study ending prematurely and the limited data available, the confidence interval was not reported. This data is NOT available as it was never provided to GTx- the median was the only reported value. Due to the study ending prematurely and the limited data available, the confidence interval was never provided to GTx- the median was the only reported value. All good cause efforts to locate the data have been exhausted, data are missing and hence not available to be reported.

6. Secondary Outcome: Time to Progression in All Subjects
Description: To estimate the time to progression in subjects receiving Gtx-024 9 mg and 18 mg in all subjects. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Time to progression was assessed up through 24 months.
Time Frame: From randomization to tumor progression or death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GTx-024 9 mg | GTx-024 18 mg
Number analyzed (Participants) | 72 | 64
months | 5.3 [NA to NA] — Due to the study ending prematurely and the limited data available, the confidence interval was not reported. This data is NOT available as it was never provided to GTx- the median was the only reported value. All good cause efforts to locate the data have been exhausted, data are missing and hence not available to be reported. | 2.9 [NA to NA] — Due to the study ending prematurely and the limited data available, the confidence interval was not reported. This data is NOT available as it was never provided to GTx- the median was the only reported value. All good cause efforts to locate the data have been exhausted, data are missing and hence not available to be reported.

7. Other Pre Specified Outcome: Number Subjects Experiencing Adverse Events
Description: To describe the safety profile of GTx-024 9 mg and 18 mg in all subjects randomized and treated. Reported adverse events were described by system organ class (SOC) as opposed to individual events
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | GTx-024 9 mg | GTx-024 18 mg
Number analyzed (Participants) | 72 | 64
Participants | 71 | 56

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | GTx-024 9 mg | GTx-024 18 mg
All-Cause Mortality (participants affected / at risk) | 8/72 | 8/64
Serious Adverse Events (participants affected / at risk) | 6/72 | 10/64
Other Adverse Events (participants affected / at risk) | 71/72 | 56/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GTx-024 9 mg (N=72) | GTx-024 18 mg (N=64)
diabetes (Endocrine disorders) | 1 | 0
hypercalcemia (Investigations) | 1 | 4
increased serum creatinine (Investigations) | 0 | 1
acute kidney failure (Renal and urinary disorders) | 1 | 1
cardiac failure (Cardiac disorders) | 0 | 2
anemia and marrow failure (Blood and lymphatic system disorders) | 0 | 1
sepsis (Infections and infestations) | 2 | 2
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
increased AST (Investigations) | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 0
pain (Musculoskeletal and connective tissue disorders) | 1 | 1
cellulitis (Infections and infestations) | 1 | 0
pneumonia (Infections and infestations) | 0 | 1
gastritis (Gastrointestinal disorders) | 0 | 1
hypertension (Cardiac disorders) | 1 | 1
myocardial infarction (Cardiac disorders) | 0 | 1
h pylori infection (Infections and infestations) | 0 | 1
tumor flare (Investigations) | 0 | 2
pyrexia (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GTx-024 9 mg (N=72) | GTx-024 18 mg (N=64)
GI disorder (Gastrointestinal disorders) | 25 | 18
general disorder (General disorders) | 25 | 12
investigations (Investigations) | 17 | 15
musculoskeletal (Musculoskeletal and connective tissue disorders) | 11 | 12
metabolism (Metabolism and nutrition disorders) | 8 | 11
nervous system (Nervous system disorders) | 10 | 7
skin (Skin and subcutaneous tissue disorders) | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT02463032/Prot_SAP_000.pdf